CLINICAL TRIAL: NCT06981117
Title: Jockey Club Stand-by-U Caregivers Community Support Project
Brief Title: Jockey Club Stand-by-U Caregivers Community Support Project: In-home Respite for Caregivers of Older Adults
Acronym: StandByU2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0048-007; 2024-0048-007 (Other Grant/Funding Number: The Hong Kong Jockey Club Charities Trust)
Record Dates: First submitted 2025-05-08; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Caregiver Burnout; Caregiver Wellbeing
Keywords: caregiver; caregiving burden; caregiver wellbeing
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caregivers - Mild Needs (Experimental): Caregivers in Mild Needs level will receive 12 hours of respite service within 3 months
  Interventions: Other: 12 hr Respite Service
- Caregivers - Moderate Needs (Experimental): Caregivers in Moderate Needs level will receive 36 hours of respite service within 3 months
  Interventions: Other: 36 hr Respite Service
- Control Group (No Intervention): Control Group will receive no service.

INTERVENTIONS:
Other: 12 hr Respite Service — 12 hours of respite service within 3 months will be provided by volunteers. Volunteers will provide elderly-sitting service (accompany the care recipient) during the service session, and provide cognitive training or physical training to the care recipient if situation allows.
  Arms: Caregivers - Mild Needs
Other: 36 hr Respite Service — 36 hours of respite service within 3 months will be provided by substitute caregivers. Substitute caregivers will provide elderly-sitting service (accompany the care recipient) during the service session, and provide cognitive training or physical training to the care recipient if situation allows.
  Arms: Caregivers - Moderate Needs

SUMMARY:
The goal of this study is to investigate whether the in-home respite service model is effective in relieving caregiver's burden and improving their mental wellbeing. Caregivers are triaged into four levels of needs using a self-developed screening tool. Those screened as mild and moderate levels are admitted to the study, while those in low or high-needs levels are referred to other services.

Caregivers admitted in this study will receive either 12 or 36 hours of in-home respite services as the intervention. Trained volunteers or substitute caregivers will visit their home to take care the older adults, providing several hours of free time for the caregivers.

Assessments are conducted before and immediate after the intervention, and 3, 6, 12 months after the completion of intervention, to measure the changes in mental wellbeing of the caregivers.

A control group with no respite service provided is recruited to compare the effects in the changes of mental wellbeing.

DETAILED DESCRIPTION:
All participants will provide informed consent at the time of enrolment. Both caregivers and their care recipients will complete assessment before the respite service period.

Care recipients are assessed for their self-dependent ability in daily activities and their physical health condition.

Caregivers are screened for their overall needs level using a self-developed multidimensional screening tool. Those screened as High Needs level will be referred professional services. Those screened as Low will be recommended to join centre-based services. Caregivers who are in Mild or Moderate needs levels will be admitted to this project. They are also assessed using standard tests for measuring changes in mental health (using Depression Anxiety Stress Scales - Short Form (DASS-21)), caregiving burden (using Chinese Version of the Zarit Caregiver Burden Interview) and quality of life (using EQ-5D-5L).

As the intervention, caregivers in Mild-needs level will receive 12 hours of in-home respite service, whereas those in Moderate-level will receive 36 hours of service. Volunteer or substitute caregivers will provide in-home elderly-sitting service so that the caregivers can have some private time for themselves.

At the end of the intervention, caregivers and care recipients will complete the assessment again to measure the changes of their physical and mental health.

All participants will be contacted again for follow-up assessment 3, 6 and 12 months after the completion of intervention.

A control group with no respite service provided is recruited to compare the effects in the changes of mental wellbeing. They are contacted 3, 6 and 12 months after baseline measurement.

ELIGIBILITY:
Caregivers and Control group

Inclusion Criteria:

* aged 18 or above
* provide care to at least one homebound older adult (aged 60 or above)
* provide no less than 6 hours of caregiving per week
* able to communicate in either Cantonese, Mandarin or English

Exclusion Criteria:

* Care recipient is receiving long-term care service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5166 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score in caregiving needs measured by Multidimensional screening tool after the intervention | Baseline and Immediate after intervention
  The Multidimensional screening tool is a self-developed tool that measures different aspects of caregiving needs over the past 1 week period. It is a 22-item scale, with 8 items that determines the overall needs level and the others for four aspects of needs: physical health, mental health, social support and care needs. Possible score is from 8 to 32 with lower score indicates lower caregivers' needs.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in mental wellbeing measured by DASS-21 scale after intervention | Baseline and Immediate after intervention
  The DASS-21 comprises 21 items that assess symptoms of depression, anxiety, and stress over the past week. Each item is rated on a 4-point Likert scale, with higher scores indicating greater symptom severity. The total scores for each subscale (Depression, Anxiety, Stress) are calculated by summing the relevant item scores. Possible score for each subscale ranged from 0 to 42, with 0 indicates best outcome and 42 the worst outcome.
  Reductions in DASS-21 scores indicate improvements in symptoms of depression, anxiety, and stress following the intervention.
  Change in score = Immediate after intervention- baseline
Change in score from baseline in caregiving burden measured by CZBI after intervention | Baseline and Immediate after intervention
  The Chinese version of Zarit Caregiver Burden Inventory (CZBI) is a widely used tool designed to assess caregiver burden and distress experienced by individuals caring for a loved one with a chronic illness or disability. It comprises of 12 items, and each item is rated on a 5-point Likert scale. Possible score ranged from 0 to 48, with higher scores indicating greater levels of caregiver burden.
  Change in score= Immediate after intervention - baseline
Change in score from baseline in quality of life measured by EQ-5D-5L after intervention | Baseline and Immediate after intervention
  The EQ-5D-5L is a standardized instrument used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses are converted into a single index value representing overall health status using Hong Kong's normative value. The primary outcome measure in this study is the change in EQ-5D-5L index scores from baseline to post-intervention/follow-up assessments. 1 equals to perfect health and more negative numbers indicates worse health.
  Change in health index = Immediate after intervention - baseline
Retention of changes of Primary outcome 1 to 4 after the end of intervention | Baseline, immediate after service, 3, 6 and 12 months after the intervention
  Caregivers will complete the primary outcome measurements (1 to 4) again 3, 6 and 12 months after the end of the intervention. They will not receive any in-home respite service from the project in between the measurement periods.
  Changes in score of each scale in Primary Outcome 1 to 4 will be measured. Participants with improved/sustained score indicates better retention.

OTHER OUTCOMES:
Respite service details in each session, including the duration and content | After each respite session
  Volunteer and Substitute Caregivers will provide a service record after each respite session, detailing the activities in each session and any potential problems observed.
  Measurements include the time of each respite session and the type of activities the caregivers and care recipient do in each session.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Weiqun Lou, Principal Investigator — The University of Hong Kong
Locations (1):
- Sau Po Centre on Ageing, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol will be published and avaliable for public. Informed consent form and anonymous data will be uploaded to HKU Data Repository under embargo protection.
Access Criteria: Study protocol will be open to public. Informed consent form and anonymous data will be uploaded to HKU Data Repository under embargo protection, and will be provided under request.

REFERENCES:
- [Derived] Hui NY, Wang LD, Yiu J, Feng MG, Lu P, Lou VWQ. JC Stand-by-U- development and evaluation of an in-home respite service model using mixed-method quasi-experimental design: study protocol. BMC Geriatr. 2025 Aug 27;25(1):665. doi: 10.1186/s12877-025-06294-w. PMID 40866876